CLINICAL TRIAL: NCT00170326
Title: Progressive Ventricular Dysfunction Prevention in Pacemaker Patients
Acronym: Prevent-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PreVent-HF
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2025-07-03 (Actual); Status verified 2017-04

CONDITIONS: Cardiac Pacing Indication classI/IIa According AHA/ACC
Keywords: Permanent Pacing artificial internal

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Video tapes are provided by the central study organization and are labelled by numbers. The tapes are sent to the echocardiography core laboratory (Malaga, Spain) and are read by the Director of the Echo Core Lab (J.J. Gomez-Doblas). The echo examiner is blinded as to the point of time of the recording and assignment of treatment, although the presence of a LV lead may be adumbrated by visible artefacts.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dual Chamber pacing (Active Comparator): conventional dual-chamber pacemaker/ICD implantation with the ventricular lead in the right ventricular apex
  Interventions: Procedure: dual-chamber pacemaker implantation
- Biventricular pacing (Experimental): Biventricular pacing: dual-chamber biventricular pacemaker/ICD implantation with leads at the right ventricular apex and the left ventricle
  Interventions: Procedure: biventricular dual-chamber pacemaker implant

INTERVENTIONS:
Procedure: dual-chamber pacemaker implantation — Dual Chamber pacing via conventional DDD(R) right ventricular pacemaker or in case of ICD indication a standard dualchamber ICD device.
  Other Names: DDD pacing, RV
  Arms: Dual Chamber pacing
Procedure: biventricular dual-chamber pacemaker implant — Biventricular pacemaker system or in case in ICD indication a BIV ICD
  Other Names: InSync 8040, InSync III 8042
  Arms: Biventricular pacing

SUMMARY:
The purpose of this pilot study is to evaluate the progression of ventricular dysfunction in patients with ventricular dysfunction within the permanent pacing population.

DETAILED DESCRIPTION:
The interventricular synchrony is one of the components of a proper cardiac function. When there is no synchrony -as in left bundle block (LBBB)- the clinic consequences should have little importance in patients with a healthy heart or a great importance in patients suffering heart failure (HF), specially in those with severe grade of HF, the benefit of cardiac resynchronization by pacing both ventricles or left ventricle (LV)should means healthy improvement in patients. All previous studies done in HF, are in patients with symptomatic HF. The importance of stop progression of latent HF in patients with asymptomatic ventricular dysfunction (VD)in permanent pacing indication patients. Pacing may accelerate HF progression by dissincronyzing ventricles. ACE inhibitors studies in asymptomatic VD gave positive results.

The PreVent-HF is an international, multicenter, prospective, randomized, single-blinded pilot trial specifically designed to evaluate as main objective the progression of VD in permanent pacing population.

ELIGIBILITY:
Inclusion Criteria:

* Meet Class I and/or Class IIa implantation criteria for permanent cardiac pacing according to the guidelines given by the American College of Cardiology (ACC)/American Heart Association(AHA).

Exclusion Criteria:

* Expected ventricle stimulation <80% of the time
* Impossibility of dual chamber stimulation in the absence of AF
* Severe heart failure (NYHA Functional class III-IV) previous to indication for pacing device implant
* Patient needs revascularization within 3 months
* Myocardial infarction in the last 3 months
* Cardiac surgery performed in the last 3 months
* Hypertrophic cardiomyopathy
* Constrictive pericarditis
* Bad echo window
* Previous system implanted (ICD or pacemaker)
* Aortic stenosis
* Patient has a mechanical right heart valve
* Patient <18 years
* Pregnancy
* Patient has medical conditions that would preclude the testing required by the protocol, or limit study participation
* Life expectancy <1year
* Patient is unwilling or unable to cooperate or give written informed consent.
* Patient is or will be inaccessible for follow-up at the study center.
* Patients who are participating or planning to participate in other clinical trials during the clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2002-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Evolution of the ejection fraction (EF) of the left ventricle (LV) and the ventricular volumes. | 12 months

SECONDARY OUTCOMES:
Combined endpoint of cardiac mortality, appearance of HF and hospitalization due to cardiovascular problems. Morbidity. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo De Teresa, MD, Principal Investigator — Hospital Clínico Universitario Virgen de la Victoria, Málaga, Spain; Javier Alzueta, MD, Principal Investigator — Hospital Clinico Universitario Virgen de la Victoria, Málaga, Spain; Ignacio Fernández Lozano, MD, Principal Investigator — Hospital Puerta de Hierro, Madrid, Spain; Juan José Gómez Doblas, MD, Principal Investigator — Hospital Clínico Universitario Virgen de la Victoria, Málaga, Spain; Francisco Navarro López, MD, Principal Investigator — Hospital Clinic i Provincial, Barcelona, Spain; A. Curnis, MD, Principal Investigator — Ospedale Civile Brescia, Italy; Xavier Navarro Michel, MD, Principal Investigator — Medtronic Ibérica, S.A., Barcelona, Spain; M. Stockburger, MD, Principal Investigator — Charite, Campus Virchow-Klinikum, Berlin, Germany; Gervasio Lamas, MD, Principal Investigator — Mount Sinai Clinical Center, Miami, FL, USA
Locations (5):
- Spain (5):
  - Hospital General de Alicante, Alicante
  - H. Infanta Cristina, Badajoz
  - H. Clínic i Provincial, Barcelona
  - H. Puerta de Hierro, Madrid
  - H. C. U. Virgen de la Victoria, Málaga

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Teresa E, Gomez-Doblas JJ, Lamas G, Alzueta J, Fernandez-Lozano I, Cobo E, Navarro X, Navarro-Lopez F, Stockburger M. Preventing ventricular dysfunction in pacemaker patients without advanced heart failure: rationale and design of the PREVENT-HF study. Europace. 2007 Jun;9(6):442-6. doi: 10.1093/europace/eum064. Epub 2007 Apr 25. PMID 17460018
- [Result] Stockburger M, Gomez-Doblas JJ, Lamas G, Alzueta J, Fernandez-Lozano I, Cobo E, Wiegand U, Concha JF, Navarro X, Navarro-Lopez F, de Teresa E. Preventing ventricular dysfunction in pacemaker patients without advanced heart failure: results from a multicentre international randomized trial (PREVENT-HF). Eur J Heart Fail. 2011 Jun;13(6):633-41. doi: 10.1093/eurjhf/hfr041. PMID 21613427
- [Result] Stockburger M, de Teresa E, Lamas G, Desaga M, Koenig C, Habedank D, Cobo E, Navarro X, Wiegand U. Exercise capacity and N-terminal pro-brain natriuretic peptide levels with biventricular vs. right ventricular pacing for atrioventricular block: results from the PREVENT-HF German Substudy. Europace. 2014 Jan;16(1):63-70. doi: 10.1093/europace/eut217. Epub 2013 Jul 16. PMID 23861381